CLINICAL TRIAL: NCT07005752
Title: Multi-center, Randomized, Double-blind, Active Controlled, Parallel Clinical Trial for the Evaluation of the Efficacy and Safety of CnU Cap. 750 mg in Patients With Cholesterol Gallstone
Brief Title: A Study to Evaluate the Efficacy and Safety of CnU Capsule 750 mg in Patients With Cholesterol Gallstones(GB Stones).
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Myungmoon Pharma. Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MMP-401
Record Dates: First submitted 2025-05-14; First posted 2025-06-05 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cholesterol Cholelithiasis
Keywords: Cholesterol gallstone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CnU capsule 250 mg(1 capsule) and Ursa placebo tablet 200 mg(1 tablet) (Experimental)
  Interventions: Drug: CnU cap. 250mg & Ursa placebo tab. 200mg
- Ursa tablet 200 mg(1 tablet) and CnU placebo capsule 250 mg(1 capsule) (Active Comparator)
  Interventions: Drug: Ursa tab. 200mg & CnU placebo cap. 250mg

INTERVENTIONS:
Drug: CnU cap. 250mg & Ursa placebo tab. 200mg — CnU capsule(Magnesium Salt Trihydrate of Chenodeoxycholic Acid and Ursodeoxycholic Acid) and Ursa placebo tablet will be orally administered three times a day after meals at regular intervals for a total of 24 weeks.
  Arms: CnU capsule 250 mg(1 capsule) and Ursa placebo tablet 200 mg(1 tablet)
Drug: Ursa tab. 200mg & CnU placebo cap. 250mg — Ursa tablet(Ursodeoxycholic Acid) and CnU placebo capsule will be orally administered three times a day after meals at regular intervals for a total of 24 weeks.
  Arms: Ursa tablet 200 mg(1 tablet) and CnU placebo capsule 250 mg(1 capsule)

SUMMARY:
The objective of this clinical trial is to evaluate the efficacy and safety of CnU capsule 750 mg administration in patients with Cholesterol gallstone (radiolucent gallstones)

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have voluntarily agreed to participate in this clinical trial
2. Adults aged 19 years and older
3. Individuals diagnosed with gall bladder stone(GB stone) with a maximum diameter size of 15 mm or less, as determined by abdominal ultrasonography at the screening stage, and who have radiolucent GB stones on plain abdominal X-ray

Exclusion Criteria:

1. Medical History

1. Patients with frequent biliary colic or biliary infections (severe pancreatic changes, such as ileal resection, resection surgery, or partial ileitis, may alter the composition of bile acids circulating in the intestines).
2. Patients with obstructive jaundice.
3. Patients with liver disease.
4. Patients with severe kidney disease.
5. Patients with severe biliary obstruction (due to choleretic effects, symptoms may worsen).
6. Patients with underlying diseases that could worsen biliary obstruction (such as biliary cancer, cholangitis, or biliary cysts).
7. Patients with acute cholecystitis.
8. Patients with peptic ulcers (due to mucosal irritation, symptoms may worsen).
9. Patients with inflammatory bowel diseases, such as Crohn's disease.
10. Patients with cholestasis.
11. Patients with abnormal gallbladder contraction.
12. Individuals with a history of malignant tumors within 5 years prior to the screening stage.
13. Individuals with a history of gastrointestinal surgery.
14. Individuals known to have hypersensitivity to the ingredients or additives of the clinical trial drug.
15. Individuals showing clinically significant disorders in the cardiovascular, gastrointestinal, respiratory, endocrine, or central nervous systems, or individuals who have had or currently have a mental disorder that could significantly affect this clinical trial.
16. Individuals with drug or alcohol addiction.
17. Individuals with genetic disorders such as galactose intolerance, Lapp lactase deficiency, or glucose-galactose malabsorption.

2. Individuals showing abnormal test results at the screening stage:

1. BMI ≥ 35 kg/m².
2. ALT or AST > 2.0 x ULN.
3. Total bilirubin > 2.0 x ULN.
4. eGFR < 60 mL/min/1.73 m² (CKD-EPI formula).
5. Positive results in serum tests (HBsAg, HCV Ab, HIV Ab, Syphilis reagin test).

3. Contraindicated drugs and therapies

The following drugs may be used after a washout period and registration:

1. Medications that increase bile secretion within 1 week prior to screening (e.g., estrogen, hormonal contraceptives, some lipid-lowering agents), or medications that reduce blood cholesterol (e.g., clofibrate).
2. Medications containing cholestyramine, colestipol, activated charcoal, magnesium, or aluminum hydroxide antacids within 2 weeks prior to screening.
3. Oral bile acid dissolution agents within 4 weeks prior to screening (e.g., chenodeoxycholic acid (CDCA), ursodeoxycholic acid (UDCA), HMG-CoA reductase inhibitors, Terpene).
4. Oral anti-diabetic medications (e.g., tolbutamide).
5. Individuals who have received bile acid treatment within 4 weeks prior to screening.

The following drugs cannot be used regardless of the washout period: Alpha-methyldopa.

4. Pregnant and breastfeeding women

5. Contraception

Participants and their spouses (or partners) who do not use medically acceptable contraceptive methods throughout the clinical trial period:

1. Use of intrauterine devices (IUD) or intrauterine systems (IUS) with proven failure rates of pregnancy.
2. Use of dual barrier contraception (male condom and cervical cap: contraceptive vaginal diaphragm or cervical cap) combined with spermicides.
3. Sterilization procedures (vasectomy, tubal ligation or cauterization, hysterectomy).

6. Other individuals deemed inappropriate for participation in the clinical trial by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Response to dissolution therapy | From baseline to the end of treatment at 24 weeks
  Response to dissolution therapy at 24 weeks compared to baseline in patients with Cholesterol gallstones.
  The dissolution response rate is defined as the sum of the GB stones complete and partial dissolution rates.

SECONDARY OUTCOMES:
1) GB stones complete dissolution rate 2) GB stones partial dissolution rate 3) GB stones dissolution rate | From baseline to the end of treatment at 24 weeks
  1. GB stones complete dissolution rate: The complete GB stones dissolution rate is defined as the proportion of subjects with no detectable gallbladder stones on ultrasonography.
  2. GB stones partial dissolution rate: The partial GB stones dissolution rate is defined as the proportion of subjects who show a reduction of more than 50% in GB stones volume.
  3. GB stones dissolution rate: The GB stones dissolution rates are defined as the rate of reduction in GB stones volume and the area of gallbladder sludge as measured by ultrasonography.

CONTACTS AND LOCATIONS:
Locations (6):
- South Korea (6):
  - Pusan National University Hospital, Busan
  - CHA Bundang Medical Center, Gyeonggi-do
  - Hallym University Dongtan Sacred Heart Hospital, Gyeonggi-do
  - Soonchunhyang University Cheonan Hospital, Gyeonggi-do
  - Inha University Hospital, Incheon
  - Gangnam Severance Hospital, Seoul